CLINICAL TRIAL: NCT04199494
Title: Antibiotic Stewardship Program in Pancreatic Surgery: a Multicenter Time Series Analysis (BIOSTEPS).
Acronym: BIOSTEPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Sponsor
Other Study IDs: TRS 2018-00001695
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-12

CONDITIONS: Surgical Site Infection; Antibiotic Resistant Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Antibiotic Stewardship Program — The patient do the routinely preoperative lab tests, including the rectal swab (RS). The Antibiotic Stewardship Program (ASP) has been shown to effectively reduce unnecessary antibiotic use and optimize the treatment of infectious diseases. To be successful, multiple aspects should be considered in the ASP. Initially, the infection control specialists will follow the routine activity of each department in order to define what could immediately be improved. Internal antibiotic prophylaxis and therapy guidelines will be defined and shared between groups. The RS, collected at the preoperative testing, is evaluated by the infection control specialist. In case of identification of MDR bacteria, each patient will receive a tailored AP based on the antibiograms of the RS. In any case, the infection control specialist will choose the best solution for the patient avoiding the key antibiotics

SUMMARY:
Rationale: Surgical site infection (SSI) is one of the most frequently reported postoperative complication, occurring in up to one-third of patients. Its development causes a substantial increase in the clinical and economic burden of pancreatic surgery. Nowadays, the primary goal of a surgical department is the reduction of the SSI rate, based on a cautious approach to the prescription of the antibiotic prophylaxis (AP) to avoid the spread of multi-drug resistant (MDR) bacteria. An antimicrobial stewardship program and a patient-tailored antibiotic prophylaxis could be an optimal strategy to reduce the impact of infectious complications after pancreatic surgery. However, few data are available regarding this topic.

Objective: To evaluate the useful of an antimicrobial stewardship program and a patient-tailored antibiotic prophylaxis in the reduction of the occurrence of SSI and the inappropriate use of key antibiotics in patients undergoing pancreatic surgery.

Study design: A time series study will be conducted. The antimicrobial stewardship program is shared between three national high-volume centers of pancreatic surgery. Statistical significance and effect size were calculated by segmented regression analysis of interrupted time series of drug use, SSI rate, and costs for 3 years before and after the introduction of the program.

Study population: Patients with an indication for elective pancreatic surgery.

Main study parameters/endpoints: Primary outcome is the reduction of SSI rate. Secondary outcomes are the reduction of the use of the key antibiotics (such as piperacillin/tazobactam and carbapenems), the microbial whole-genome sequencing (WGS) of the carbapenemase-producing Enterobacteriaceae, and the reduction of the treatment costs

DETAILED DESCRIPTION:
A multicenter time series with segmented regression analysis will be conducted at three national high-volume centers of pancreatic surgery: The General and Pancreatic Surgery Department, Pancreas Institute, of Verona, the Oncological and Robotic General Surgery, Careggi University of Florence, and the Department of Surgery, University Campus Bio-Medico of Rome. All patients visited at the General and Pancreatic Surgery Department, Pancreas Institute, of Verona, the Oncological and Robotic General Surgery, Careggi Hospital, University of Florence, and the Department of Surgery, University Campus Bio-Medico of Rome and scheduled for pancreatic resection will be enrolled. The patients will be submitted to the routinely diagnostic preoperative procedures, including the RS culture, two weeks before surgery. All patients enrolled will receive a preoperative clinical visit two weeks before surgery. During the patient's interview, the surgeon will collect the medical history, exposing the clinical and surgical perioperative pathways. The patient is also submitted to the routinely preoperative lab tests, including the RS. The study design is based on evidence collected by previous studies of the group and after a systematic review of the literature. The ASP has been shown to effectively reduce unnecessary antibiotic use and optimize the treatment of infectious diseases. To be successful, multiple aspects should be considered in the ASP. Initially, the infection control specialists will follow the routine activity of each department in order to define what could immediately be improved. Internal antibiotic prophylaxis and therapy guidelines will be defined and shared between groups. The RS, collected at the preoperative testing, is evaluated by the infection control specialist. In case of identification of MDR bacteria, each patient will receive a tailored AP based on the antibiograms of the RS. In any case, the infection control specialist will choose the best solution for the patient avoiding the key antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective pancreatic resection
* Age ≥ 18 years
* American Society of Anesthesiologists (ASA) score < 4
* The ability of the subject to understand the character and individual consequences of the clinical trial
* Written informed consent

Exclusion Criteria:

* Under 18 years of age
* ASA score ≥4
* Immune suppressed patients
* Pregnant women
* Participation in another study with interference of study outcomes
* Impaired mental state or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients visited at the General and Pancreatic Surgery Department, Pancreas Institute, of Verona, the Oncological and Robotic General Surgery, Careggi Hospital, University of Florence, and the Department of Surgery, University Campus Bio-Medico of Rome and scheduled for pancreatic resection will be enrolled. The patients will be submitted to the routinely diagnostic preoperative procedures, including the Rectal Swab culture, two weeks before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-16 (Estimated)

PRIMARY OUTCOMES:
SSI rate after pancreatic surgery | 30th day after surgery
  To evaluate the useful of an antimicrobial stewardship program and a patient-tailored antibiotic prophylaxis in the reduction of the occurrence of SSI until 30th day after surgery in patients undergoing pancreatic surgery

SECONDARY OUTCOMES:
Antibiotic Stewardship Program in Pancreatic Surgery | 30th day after surgery
  To evaluate the useful of an antibiotic stewardship program in the change of the inappropriate use of key antibiotics, such as piperacillin/tazobactam and carbapenems, in administered for prophylaxis or treatment of the SSI
Whole genome sequencing of MDR bacteria | 30th day after surgery
  To analyze the genotype of the carbapenemase-producing Enterobacteriaceae performing the microbial WGS
Treatment costs | 30th day after surgery
  To evaluate the useful of an antibiotic stewardship program in the change of the treatment costs

CONTACTS AND LOCATIONS:
Locations (1):
- AOUI Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No